CLINICAL TRIAL: NCT06868199
Title: A Phase I/II, First-in-Human (FIH), Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LM-168 as a Single Agent or in Combination With Toripalimab in Subjects With Advanced Solid Tumours
Brief Title: A Study of LM-168 as a Single Agent or in Combination With Toripalimab in Subjects With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM168-01-101
Record Dates: First submitted 2025-02-06; First posted 2025-03-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumours
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- LM-168 Dose Escalation (Experimental)
  Interventions: Drug: LM-168
- LM-168 Dose Expansion (Experimental)
  Interventions: Drug: LM-168
- LM-168 combination dose escalation (Experimental)
  Interventions: Drug: LM-168; Drug: Toripalimab
- LM-168 combination dose expansion (Experimental)
  Interventions: Drug: LM-168; Drug: Toripalimab

INTERVENTIONS:
Drug: LM-168 — Q3W,Intravenous Drip
Drug: Toripalimab — Q3W,Intravenous
  Arms: LM-168 combination dose escalation; LM-168 combination dose expansion

SUMMARY:
For phase I ,this study is to assess the safety and tolerability, obtain the recommended phase 2 dose (RP2D) and/or Maximum Tolerated Dose (MTD) for LM-168 as a single agent or in combination with toripalimab in subjects with advanced solid tumours.

For phase II ,this study is to assess the preliminary anti-tumour activity of LM-168 as a single agent or in combination with toripalimab measured by objective response rate (ORR) in subjects with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Aged ≥18 years old (including boundary values) , male or female.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancy ≥ 3 months.
5. In dose escalation stage, subjects must have histological or cytological confirmation of recurrent or refractory advanced solid tumours, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
6. In dose expansion stage, subjects must have histological or cytological confirmation of selected advanced solid tumors.
7. Pre-treatment archived tumour tissue or on-treatment tumour biopsy could be provided for biomarker analysis optionally.
8. At least one measurable disease.
9. Subjects must show appropriate organ and marrow function in laboratory examinations within 7 days prior to the first dose.
10. Subjects who are able to communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Participate in any other clinical trial within 28 days prior to 1st dosing of LM-168.
2. Having received prior anti-CTLA-4 or any other immunotherapy or immune-oncology (IO) agent within 28 days of commencing treatment with LM-168 or experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
3. Subjects who have received the anti-tumor treatments within the specified time periods prior to the first dosing of LM-168.
4. Any adverse event from prior anti-tumour therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
5. Subjects with uncontrolled tumour-related pain.
6. Subjects with known central nervous system (CNS) or meningeal metastasis.
7. Subjects who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
8. Subjects with esophageal or gastric varices requiring immediate intervention, or those with a history of variceal bleeding.
9. Hepatic encephalopathy, hepatorenal syndrome, Child-Pugh class B or more severe liver cirrhosis.
10. Tumor invasion of surrounding vital organs or a risk of developing esophagotracheal fistula or esophagopleural fistula.
11. Patients with a history of active or previously confirmed inflammatory bowel disease.
12. Subjects who experienced grade 3 or higher hypersensitivity to the treatment that contains monoclonal antibody.
13. Subjects who previously experienced grade ≥ 3 immune-related adverse events during immunotherapy, as well as subjects who discontinued prior immunotherapy due to severe or life-threatening immune-related adverse events.
14. Subjects who take systemic corticosteroids (> 10 mg daily prednisone equivalents) or other systemic immunosuppressive medications within 2 weeks prior to the first dosing of LM-168.
15. Subjects with the known history of autoimmune disease.
16. Subjects with the history of idiopathic pulmonary fibrosis, organizing pneumonia , drug-induced pneumonitis, idiopathic pneumonitis, interstitial lung disease, severe radiation pneumonitis or evidence of active pneumonitis on screening chest CT scan.
17. Use of any live attenuated vaccines within 28 days prior to 1st dosing of LM-168.
18. Current or recent use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
19. Current unstable of full-dose oral or parenteral anticoagulants or thrombolytic agents for > 2 weeks prior to the first dose of LM-168.
20. Subjects who received major surgery or interventional treatment within 28 days prior to 1st dosing of LM-168 (excluding tumour biopsy, puncture, etc.).
21. Subjects who have severe cardiovascular disease.
22. Subjects who have uncontrolled or severe illness.
23. Subjects who have a history of immunodeficiency disease.
24. HIV infection, active infection including tuberculosis, HBV and HCV infection.
25. Subjects with a history of other malignancies within 5 years prior to the first administration of the study drug.
26. Child-bearing potential female who have positive results in pregnancy test or are lactating.
27. Subjects who have psychiatric illness or disorders that may preclude study compliance.
28. Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 78 weeks
  Phase I
Incidence of dose-limitingtoxicity (DLT) | 78 weeks
  Phase I
Incidence of serious adverse event (SAE) | 78 weeks
  Phase I
Temperature (Celsius) | 78 weeks
  Phase I
Pulse in BPM(Beat per Minute) | 78 weeks
  Phase I
Blood Pressure in mmHg | 78 weeks
  Phase I
Weight in Kg | 78 weeks
  Phase I
Height in centimeter | 78 weeks
  Phase I
Blood Routine examination | 78 weeks
  Phase I
Urine Routine test | 78 weeks
  Phase I
Blood biochemistry test | 78 weeks
  Phase I
Coangulation function test | 78 weeks
  Phase I
Thyroid function test | 78 weeks
  Phase I
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in HR | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in RR | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in PR | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in QRS | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in QT | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in QTcF | 78 weeks
  Phase I
ECOG(Eastern Cooperative Oncology Group) score | 78 weeks
  Phase I
Objective Response Rate (ORR) | From 78th week to 130th week (52 weeks in total)
  Phase II

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 78 weeks
  Phase I
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) | 130 weeks
  Phase I/II
PK Parameter:Time of Maximum Observed Concentration (Tmax) | 130 weeks
  Phase I/II
PK Parameter: Area Under the Concentration-time Curve(AUC) | 130 weeks
  Phase I/II
PK Parameter: Steady State Maximum Concentration(Cmax,ss) PK Parameter: Steady State Maximum Concentration(Cmax,ss) | 130 weeks
  Phase I/II
PK Parameter: Steady State Minimum Concentration(Cmin,ss) | 130 weeks
  Phase I/II
PK Parameter: Systemic Clearance at Steady State (CLss) | 130 weeks
  Phase I/II
PK Parameter: Accumulation Ratio (Rac) | 130 weeks
  Phase I/II
PK Parameter: Elimination Half-life (t1/2) | 130 weeks
  Phase I/II
PK Parameter: Volume of Distribution at Steady-State (Vss) | 130 weeks
  Phase I/II
PK Parameter: Degree of Fluctuation (DF) | 130 weeks
  Phase I/II
Immunogenicity testing | 130 weeks
  Phase I/II
Duration of Response (DOR) in Month | 130 weeks
  Phase I/II
Disease control rate (DCR) in percentage | 130 weeks
  Phase I/II
progression-free survival (PFS) in Month | 130 weeks
  Phase I/II
Changes of target lesions from baseline in Millimeter | 130 weeks
  Phase I/II
Temperature (Celsius) | From 78th week to 130th week (52 weeks in total)
  Phase II
Pulse in BPM(Beat per Minute) | From 78th week to 130th week (52 weeks in total)
  Phase II
Blood Pressure in mmHg | From 78th week to 130th week (52 weeks in total)
  Phase II
Weight in Kg | From 78th week to 130th week (52 weeks in total)
  Phase II
Height in centimeter | From 78th week to 130th week (52 weeks in total)
  Phase II
Blood Routine examination | From 78th week to 130th week (52 weeks in total)
  Phase II
Urine Routine test | From 78th week to 130th week (52 weeks in total)
  Phase II
Blood biochemistry test | From 78th week to 130th week (52 weeks in total)
  Phase II
Coangulation function test | From 78th week to 130th week (52 weeks in total)
  Phase II
Thyroid function test | From 78th week to 130th week (52 weeks in total)
  Phase II
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | From 78th week to 130th week (52 weeks in total)
  Phase II
ECOG(Eastern Cooperative Oncology Group) score | From 78th week to 130th week (52 weeks in total)
  Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Qin, Study Director — LaNova Medicines Limited
Locations (6):
- Australia (5):
  - Macquarie University, Ryde, New South Wales
  - MUPharm Pty Limited trading as Macquarie University Hospital Parmarcy, Ryde, New South Wales
  - Cancer Care Wollongong Pty Limited, Wollongong, New South Wales
  - Bayview Health-Investigational Drug Services, Perth, Western Australia
  - One Clinical Reasearch, Perth, Western Australia
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No